CLINICAL TRIAL: NCT05995886
Title: Facebook Intervention for Preventing Opioid Relapse Among American Indian Women: Wiidookaage'Win Pilot Preparatory Study (Aim 2)
Brief Title: Using Facebook to Support Opioid Recovery Among American Indian Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-005038; DA40316-08S2 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Opioid Use Disorder
Keywords: American Indian or Alaska Native; Internet-based Intervention; Community-based Participatory Research; Minnesota; Ethnic and Racial Minorities; Women's Health
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wiidookaage'win Facebook Group (Experimental): The Wiidookaage'win Facebook Group is an online, asynchronous group intervention that will run for 3-months with approximately 30 days of content developed. It is private and hidden, meaning only those in the study will be able to see or find the group. It will be moderated by two women from the study team (one AIAN and one biracial). A back-up moderator will also have access to the group. Participants will be able to comment, react, view, and post in the intervention group, and are encouraged to interact with one another.
  Interventions: Behavioral: Wiidookaage'win Facebook Group
- Online Resources Landing Page (No Intervention): The Online Resources Landing Page was developed by the study team using https://carrd.co. It includes links to local programs in family services, substance use recovery, legal advocacy, etc. which already exist and may help support their recovery.

INTERVENTIONS:
Behavioral: Wiidookaage'win Facebook Group — An online social media group program that incorporates social support, mindfulness-based, and cultural practices that may support OUD recovery.
  Arms: Wiidookaage'win Facebook Group

SUMMARY:
The purpose of this study is to find out whether a Facebook group will help Native women in recovery from opioid use.

ELIGIBILITY:
Inclusion Criteria:

1. AIAN person based on self-reported race/ethnicity
2. Gender identity as a woman
3. At least 18 years of age with no upper age limit
4. Resides in Minnesota
5. Meets criteria for OUD based on the DSM-5 Checklist (American Psychiatric Association, 2013)
6. Self-reports at least one month of abstinence from opioid use based on TLFB interview and negative urine opiate screen
7. Current use of MOUD
8. Is comfortable speaking and reading English
9. Has an existing Facebook account or willing to set one up
10. Is willing and able to participate in the Facebook intervention for 3 months
11. Has access to broadband internet on a mobile phone/computer/tablet at any location
12. Is willing and able to travel to a community clinic in Minneapolis, Minnesota for the UDS or is willing to and able to complete a virtual Zoom UDS visit.
13. Provides written informed consent

Exclusion Criteria:

1. Self-reports current suicidality based on the Concise Heath Risk Tracking scale
2. Participated in prior study phases (Aim 1 formative work) of NIDA CTN-0123

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants may be cisgender or transgender women. They may also identify as Two Spirit and include "woman" as part of their gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Facebook Intervention | 3 months
  The study team will measure the feasibility from the combined reports of recruitment, study retention, level of Facebook intervention uptake/engagement, and treatment satisfaction.

SECONDARY OUTCOMES:
Timeline Follow-back Interview and UDS to measure Opioid Abstinence | 6 months
  The study team will explore the preliminary differential impact of the intervention compared with the control condition on opioid abstinence and MOUD continuation. Opioid and other substance use will be assessed through monthly Timeline Follow-Back (TLFB) interviews (Sobell & Sobell, 1992; Wray et al., 2016). At 1, 3, and 6-months, the study team will obtain a UDS that will be used along with the TLFB interviews to measure opioid abstinence.
Reporting MOUD continuation | 6 months
  The study team will summarize MOUD continuation as the proportion of participants reporting current use at 6-month follow-up.

OTHER OUTCOMES:
Perceived Stress Scale and Communal Mastery Scale | 3 months
  The study team will explore the differential impact of the intervention compared with the control condition on constructs targeted by our intervention, specifically perceived stress and coping with stressful life circumstances from a more collectivist orientation, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20559266